CLINICAL TRIAL: NCT01194297
Title: Immune Responses in Preterm and Full-Term Infants Following Live, Attenuated Influenza Vaccination
Brief Title: Study of Live, Attenuated Influenza Vaccination in Preterm and Full-Term Infants
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Carl D'Angio, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25914
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Influenza
Keywords: influenza; premature infant; very low birth weight infant; immunization; vaccine
MeSH Terms: conditions — Influenza, Human; Premature Birth | interventions — Influenza Vaccines; FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Live attenuated influenza vaccine (Experimental): One dose of live attenuated influenza vaccine, according to routine immunization recommendations
  Interventions: Biological: Live attenuated influenza vaccine
- Inactivated influenza vaccine (Active Comparator): One dose of inactivated influenza vaccine, according to routine immunization recommendations
  Interventions: Biological: Inactivated influenza vaccine

INTERVENTIONS:
Biological: Live attenuated influenza vaccine — One dose of live attenuated influenza vaccine, according to routine immunization recommendations
  Other Names: FluMist
  Arms: Live attenuated influenza vaccine
Biological: Inactivated influenza vaccine — One dose of inactivated influenza vaccine, according to routine immunization recommendations
  Other Names: Fluzone
  Arms: Inactivated influenza vaccine

SUMMARY:
Severe influenza respiratory disease is increasingly recognized in children. Influenza hospitalization rates in high-risk infants, such as premature infants, are increased some five-fold over rates in other children. The recently-licensed live attenuated influenza vaccine (LAIV) promotes better immune responses than the trivalent inactivated vaccine, but can cause wheezing. The balance of risks and benefits for LAIV in extremely premature infants, who may be at increased risk for both influenza disease and vaccine side effects, is unknown.

The specific aim of this project is to compare the immune response and reactions of trivalent, inactivated influenza vaccine (TIV) and live, attenuated, intranasal influenza vaccine (LAIV) in groups of former premature (PT), very (V) LBW and former full-term (FT) infants aged 24-35 months.

The investigators hypothesize that the immune response in FT infants will be greater with LAIV than TIV, and that wheezing episodes will be no more than twice as frequent in LAIV as in TIV recipients.

The study will enroll 14 former premature, VLBW infants and 14 former full-term infants. Children will be randomized to receive one dose either TIV or LAIV. Vaccine reactions will be measured. One to two teaspoons mL of blood will be drawn at 0 and 7-14 days from immunization, and less than one teaspoon of blood will be drawn at 28-42 days.

DETAILED DESCRIPTION:
Background. Influenza infection causes an estimated 1 million deaths worldwide yearly. Severe influenza respiratory disease is increasingly recognized in children. Influenza hospitalization rates in high-risk infants, such as premature infants, are increased some five-fold over rates in other children. Influenza vaccine immunogenicity is generally modest even in healthy children, and influenza vaccines have been incompletely studied in premature infants. The recently-licensed live attenuated influenza vaccine (LAIV) is more immunogenic than the trivalent inactivated vaccine, but its use in infants and high risk children is limited by side effects. The risk/benefit ratio of LAIV in extremely premature infants, who may be at increased risk for both influenza disease and vaccine side effects, is unknown.

Aim. The specific aim of this project is to compare the immunogenicity and reactogenicity of trivalent, inactivated influenza vaccine (TIV) and live, attenuated, intranasal influenza vaccine (LAIV) in groups of former premature (PT), very low birth weight (VLBW) and former full-term (FT) infants aged 24-35 months.

Hypotheses.

1. The humoral immunogenicity of LAIV, as measured by hemagglutination inhibition (HI), will be greater than that of TIV. This will be the co-primary outcome for this study.
2. Vaccine reactogenicity, as measured by medically-attended wheezing episodes, will be no more than twice as frequent in LAIV as in TIV recipients. This will be the co-primary outcome for this study.
3. Functional B-cell responses, as measured by antibody secreting cell (ASC) enzyme linked immunospot (ELISPOT), will be greater in LAIV-immunized infants than TIV-immunized infants.
4. Peak T-cell cytokine responses, as measured by interferon gamma (IFNγ), interleukin (IL)-2 and IL-4 ELISPOT, will be greater in LAIV-immunized infants than TIV-immunized infants.
5. Hemagglutinin-specific nasal immunoglobulin A (IgA) will be measureable following LAIV immunization.
6. Former premature infants will have similar adaptive immune responses, but elevated reactogenicity to both vaccines, when compared to former full-term infants.

Design. The study will enroll 14 former premature, VLBW infants and 14 former full-term infants. Subjects, who will be eligible to receive either TIV or LAIV as part of routine care, will be randomized to receive one dose either TIV or LAIV, according to prevailing recommendations for influenza immunization. Randomization will be stratified by prematurity status. Vaccine reactogenicity will be measured by using parent diaries following immunization and questionnaires at each visit. Five to 10 mL of blood will be drawn at 0 and 7-14 days from immunization for isolation of peripheral blood mononuclear cells (PBMC), and 1 mL of blood will be drawn for serum separation for antibody determination at 0 and 28-42 days. Antibody levels and T- and B-cell responses to vaccine will be measured.

Potential Impact. This study is designed to assess the immunogenicity and reactogenicity of two current influenza vaccines in premature infants. The data will be used to estimate the sample size for a definitive trial in younger premature infants.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all relevant criteria (by time of influenza vaccination) to participate.

1. (a) Former premature (<32 weeks' gestation at birth), VLBW (<1500 grams' birth weight) infant, 24 months, 0 days - 35 months, 31 days of age, OR (b) Former full-term (37-42 weeks' gestation at birth), normal birth weight (>2500 grams' birth weight) infant, 24 months, 0 days - 35 months, 31 days of age.
2. Influenza immunization in prior season.
3. Eligible for either influenza immunization (TIV or LAIV).
4. Parental permission.
5. Parents likely to be able to comply with study visits.

Exclusion Criteria:

Subjects may not participate if they meet any one of these criteria.

1. Known immunodeficiency in child or in a close household contact.
2. History of:

   * Recurrent episodes of wheezing,
   * Medically-attended wheezing illness in past year, or
   * Hospitalization for a wheezing illness.
3. Systemic corticosteroid administration at time of influenza vaccination.
4. Requiring supplemental oxygen at time of influenza vaccination.
5. Contraindication to either influenza immunization (e.g. egg allergy, aspirin therapy).
6. Physician-diagnosed influenza illness in the current influenza season.
7. Any condition determined by investigator as likely to interfere with evaluation of the vaccine or be a significant potential health risk to the subject.

Ages: 24 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl T. D'Angio, MD, Principal Investigator — University of Rochester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited during influenza season 2010-2011
Pre-assignment Details: No significant pre-assignment details
Groups:
- Inactivated Influenza Vaccine: One dose of inactivated influenza vaccine, according to routine immunization recommendations
  Inactivated influenza vaccine : One dose of inactivated influenza vaccine, according to routine immunization recommendations
- Live Attenuated Influenza Vaccine: One dose of live attenuated influenza vaccine, according to routine immunization recommendations
  Live attenuated influenza vaccine : One dose of live attenuated influenza vaccine, according to routine immunization recommendations
Period: Overall Study
Arm/Group | Inactivated Influenza Vaccine | Live Attenuated Influenza Vaccine
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inactivated Influenza Vaccine | Live Attenuated Influenza Vaccine | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Humoral Immunogenicity
Description: Hemagglutinin specific antibody, as measured by hemagglutination inhibition
Time Frame: 28-42 days
Arm/Group | Inactivated Influenza Vaccine | Live Attenuated Influenza Vaccine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Medically-attended Wheezing
Description: Wheezing that triggers a visit for medical care
Time Frame: 42 days
Population: Total N
Measure: Number; unit: participants
Arm/Group | Inactivated Influenza Vaccine | Live Attenuated Influenza Vaccine
Number analyzed (Participants) | 2 | 1
participants
  wheezing | 0 | 0
  medical care | 0 | 0

ADVERSE EVENTS:
Arm/Group | Inactivated Influenza Vaccine | Live Attenuated Influenza Vaccine
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes